CLINICAL TRIAL: NCT00965237
Title: P/331/09/C: Multifocal Pilot Study: Refitting Drop Outs (GARM)
Brief Title: Multifocal Contact Lens Use in Previous Contact Lens Wearers With Near Vision Demands
Acronym: GARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-368-C-101
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2011-03-14 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifocal CL / Single vision CL + reading glasses (Other): Lotrafilcon B multifocal contact lenses (CL) worn first, with lotrafilcon B single vision contact lenses (CL) and over-reader spectacles worn second. Both contact lens products worn bilaterally on a daily wear basis; over-reader spectacles worn on an as-needed basis.
  Interventions: Device: lotrafilcon B multifocal contact lens; Device: lotrafilcon B single vision contact lens; Other: Over-reader spectacles
- Single vision CL + reading glasses / Multifocal CL (Other): Lotrafilcon B single vision contact lenses (CL) and over-reader spectacles worn first, with lotrafilcon B multifocal contact lenses (CL) worn second. Both contact lens products worn bilaterally on a daily wear basis; over-reader spectacles worn on an as-needed basis.
  Interventions: Device: lotrafilcon B multifocal contact lens; Device: lotrafilcon B single vision contact lens; Other: Over-reader spectacles

INTERVENTIONS:
Device: lotrafilcon B multifocal contact lens — Commercially marketed, silicone hydrogel, multifocal contact lens for daily wear use
Device: lotrafilcon B single vision contact lens — Commercially marketed, silicone hydrogel, single vision contact lens for daily wear use
Other: Over-reader spectacles — Reading glasses worn over single vision contact lenses for near vision work on an as-needed basis

SUMMARY:
The purpose of this study is to evaluate the use of a multifocal contact lens in people who previously wore contact lenses but discontinued due to age-related, near vision demands.

ELIGIBILITY:
Inclusion Criteria:

* has discontinued contact lens wear primarily due to age-related, near vision demands
* requires a reading add of +0.50 to +1.75 D (inclusive) and is correctable to at least 6/9 monocular, distance and near with spectacle correction
* has had an ocular examination in the last 2 years
* Other protocol-defined inclusion/exclusion criteria may apply

Exclusion Criteria:

* has any ocular disease
* has more than a 2.00D prescription difference between eyes
* cannot be fit successfully with the study contact lenses
* has any systemic disease affecting ocular health
* is using any systemic or topical medications that may affect ocular health
* has undergone corneal refractive surgery
* Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Waterloo Centre for Contact Lens Research, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Multifocal CL / Single Vision CL+ Reading Glasses: Lotrafilcon B multifocal contact lenses (CL) worn first, with lotrafilcon B single vision contact lenses (CL) and over-reader spectacles worn second. Both contact lens products worn bilaterally on a daily wear basis; over-reader spectacles worn on an as-needed basis.
Period: Period 1, One Week of Wear
Arm/Group | Multifocal CL / Single Vision CL+ Reading Glasses | Single Vision CL + Reading Glasses / Multifocal CL
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Period 2, One Week of Wear
Arm/Group | Multifocal CL / Single Vision CL+ Reading Glasses | Single Vision CL + Reading Glasses / Multifocal CL
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This reporting group includes all enrolled and dispensed subjects.
Arm/Group | Overall Study
Number analyzed (Participants) | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 48.3 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Satisfaction With the Lenses
Description: Overall satisfaction with the lenses was interpreted by and assessed by the subject as a single, retrospective measurement of one week's wear time. Overall satisfaction with the lenses was recorded on a questionnaire as a numerical rating on a scale of 1 to 100, with 1 being completely dissatisfied, and 100 being excellent, completely satisfied.
Time Frame: 1 week of wear
Population: Analysis conducted per protocol
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Lotrafilcon B Multifocal Contact Lens: Commercially marketed, lotrafilcon B, silicone hydrogel, multifocal contact lens for daily wear use
- Lotrafilcon B Single Vision Contact Lens + Reading Glasses: Commercially marketed, lotrafilcon B, silicone hydrogel, single vision contact lenses for daily wear use, with over-reader spectacles worn as needed
Arm/Group | Lotrafilcon B Multifocal Contact Lens | Lotrafilcon B Single Vision Contact Lens + Reading Glasses
Number analyzed (Participants) | 16 | 16
Units on a Scale | 82.5 (14.5) | 64.4 (22.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial. Individual subject exposure = 1 week per product, total 2 weeks.
Groups:
- Multifocal Contact Lens: Commercially marketed lotrafilcon B multifocal contact lenses
- Single Vision Contact Lens: Commercially marketed lotrafilcon B single vision contact lenses
Arm/Group | Multifocal Contact Lens | Single Vision Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No distribution of trial-specific information without express written permission of director.